CLINICAL TRIAL: NCT01947192
Title: Chlorhexidine as Coadjuvant in Dentin Adhesion of Noncarious Cervical Lesions and Failure-prognostic Variables: A Randomized Controlled Trial
Brief Title: Chlorhexidine as Coadjuvant in Dentin Adhesion of Noncarious Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Associate Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPGO0017
Record Dates: First submitted 2013-08-15; First posted 2013-09-20 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Non-carious Cervical Lesions
Keywords: Chlorhexidine; Matrix metalloproteinases (MMP) inhibitor; Adhesive system; Controlled clinical trial; Dental restoration; Noncarious cervical lesions; Dental restoration failure
MeSH Terms: interventions — Therapeutics; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Chlorhexidine (Experimental): Dentin pre-treatment with a experimental solution (chlorhexidine), after the dentin acid etching
  Interventions: Procedure: Treatment with chlorhexidine
- Water (Placebo Comparator): Application of water (placebo) after dentin acid etching.
  Interventions: Procedure: Water pre-treatment

INTERVENTIONS:
Procedure: Treatment with chlorhexidine — Application of 2% chlorhexidine digluconate (60 seconds) after the etching procedure and before the adhesive system.
  Arms: Chlorhexidine
Procedure: Water pre-treatment — Treatment of acid etched dentin with sterilized water for 60 s before adhesive system application
  Arms: Water

SUMMARY:
This study aims to evaluate the effect of chlorhexidine digluconate (CRX) application in etched dentin on the retention of noncarious cervical lesions restorations.

A randomized controlled split-mouth and blind trial will be carried out. Patients with at least two non-carious cervical lesions (NCL) will be selected. NCL will be randomly assigned according the type of teeth (incisors, canine or pre-molars) into two groups: control or experimental group (application of 2% CRX for 60 seconds after the acid etching procedure). Class V restorations will be performed out with an etch-and-rinse adhesive system (Adper Single Bond 2-3M ESPE) and a composite resin (Filtek Z350-3M ESPE) according the manufacture instructions, by previously trained operators. The restorations will be evaluated by a calibrate examiner at 1 week (baseline), and 6-month, 12-month and 24-month, using the World Dental Federation (FDI) criteria. The outcome is retention of the restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at least two non-carious cervical lesions (NCL) in anterior, canine or pre-molars;
* Patients who had more than 20 teeth in the mouth;
* Patients who were at least 18 years of age at the time of treatment and capable to understand and sign the written informed consent;
* NCL with at least 1 mm of depth in a vital permanent incisor, canine or premolar of the upper as the lower jaw.
* NCL in the facial surface of the teeth with sometimes a small part extending interproximally;
* Patients with good periodontal heath.

Exclusion Criteria:

* Patients with smoking habits, practicing bruxism, severe systemic diseases, using active orthodontic treatment, malocclusion (Angle Class II or Class III);
* Tooth with the NCL with the absent of antagonist;
* NCL wear facets upper than 50% of the incisal/occlusion surface, as a result of tooth attrition;
* Presence of caries or restorations in the area to be treated;
* Full-mouth visible plaque index (VPI) or full-mouth gingival bleeding index upper than 20%, probing depth and clinical attachment loss values exceeding 4 mm with bleeding on probing;
* Unwillingness to return for follow-ups or refuse to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Retention rates of the restoration at 24 months | 6, 12 and 24 months
  Patients will be reevaluated at each specified time point and all restoration sites will be evaluated to check if the restoration will be still in place, or if it is missing, or if there is partial retention

SECONDARY OUTCOMES:
Change from baseline in Post-operative sensitivity at 6-month | baseline and 6-month
  At each time-point, patients will be recalled and interviewed regarding any symptom related to each restorations placed.
Change from baseline in marginal staining rates at 6. 12 and 24 months | 6, 12 and 24 months
  At each time-point, patients will be recalled and restorations will be reassessed in order to record changes in the rates of marginal staining, using the World Dental Federation (FDI) criteria for restorations assessment (Hickel et al 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano Cenci, PhD, Principal Investigator — School of Dentistry-UFPel
Locations (1):
- School of Dentistry, Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774